CLINICAL TRIAL: NCT04921293
Title: Comparison Between Endogenous and Exogenous Ketosis in Patients With Non-ischemic Chronic Heart Failure With Reduced Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIE-3652-21-22-1
Record Dates: First submitted 2021-06-02; First posted 2021-06-10 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Ketosis
Keywords: Endogenous ketosis; Exogenous ketosis; Heart failure
MeSH Terms: conditions — Ketosis; Heart Failure | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Diet (Active Comparator): Standard diet incorporating current recommendations for heart failure (low sodium and liquids) and supplementation with bitter taste placebo.
  Interventions: Behavioral: Standard diet + placebo
- Endogenous Ketosis (Experimental): Ketogenic diet incorporating current recommendations for heart failure (<50gr of carbohydrates, low sodium, and liquids) for 10 days.
  Interventions: Behavioral: Ketogenic diet
- Exogenous ketosis (Experimental): Standard incorporating current recommendations for heart failure (low sodium and liquids) and supplementation with exogenous ketones (ketone monoester) for 10 days.
  Interventions: Dietary Supplement: Exogenous ketones

INTERVENTIONS:
Behavioral: Ketogenic diet — A diet with <50gr of carbohydrates per day. Monosaturated fats consumption will encourage over saturated fats
  Arms: Endogenous Ketosis
Dietary Supplement: Exogenous ketones — Administration of ketone monoester 25 ml t.i.d
  Arms: Exogenous ketosis
Behavioral: Standard diet + placebo — A standard diet incorporating current recommendations (low in sodium and low in liquids) for heart failure patients.
  Arms: Standard Diet

SUMMARY:
This randomized controlled trial will evaluate the effect of a ketogenic diet and/or exogenous administration of ketone bodies vs conventional diet on the ejection fraction of patients with non-ischemic chronic heart failure, measuring MRI biomarkers.

DETAILED DESCRIPTION:
Evidence in both animals and humans suggests ketosis could be beneficial for people living with chronic heart failure. To date, no study has compared endogenous vs exogenous ketosis in patients with chronic heart failure. We will randomize (with a 1:1:1 ratio) patients with a confirmed diagnosis of non-ischemic chronic heart failure to undergo one of the following:

1. - A ketogenic diet (<50 gr of carbohydrates per day) incorporating current recommendations for heart failure (low sodium and liquids) for 10 days.
2. - Standard diet incorporating current recommendations for heart failure (low sodium and liquids) and supplementation with exogenous ketones (ketone monoester) for 10 days.
3. - Standard diet incorporating current recommendations for heart failure (low sodium and liquids) and supplementation with bitter taste placebo.

The endpoints will be assessed using cardiac MRI and blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction <40% minimum 1 month.
* No change in optimum treatment 1 month at least.

Exclusion Criteria:

* Ischemic cardiopathy (Angio-tomography corroborated cut-point >50% obstruction, coronary angiography, or cardiac scintigraphy 6 months at least) or angina pectoris symptoms.
* Reynaud syndrome
* Metformin or SGLT-2 Inhibitors treatment, Low BMI, nutritional deficiencies.
* Creatinin clearance <30ml/min or renal replacement therapy
* MRI contraindications (prothesis, Unsupported pacemakers, claustrophobia, etc)
* Reynaud phenomenon history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Ejection fraction Improvement | 10 days
  Estimated by cardiac MRI

SECONDARY OUTCOMES:
Clinical severity | 10 days
  Estimated with the NYHA classification
Liquid retention | 10 days
  Estimated by electric bioimpedance
Blood biomarker | 10 days
  BNP

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Soto, Ph.D, MD., Principal Investigator — INCMNSZ
Locations (1):
- INCMNSZ, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Upon request to PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after publication
Access Criteria: Send email to adrian.sotom@incmnsz.mx

REFERENCES:
- [Background] Astrup A, Magkos F, Bier DM, Brenna JT, de Oliveira Otto MC, Hill JO, King JC, Mente A, Ordovas JM, Volek JS, Yusuf S, Krauss RM. Saturated Fats and Health: A Reassessment and Proposal for Food-Based Recommendations: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Aug 18;76(7):844-857. doi: 10.1016/j.jacc.2020.05.077. Epub 2020 Jun 17. PMID 32562735
- [Background] Athinarayanan SJ, Adams RN, Hallberg SJ, McKenzie AL, Bhanpuri NH, Campbell WW, Volek JS, Phinney SD, McCarter JP. Long-Term Effects of a Novel Continuous Remote Care Intervention Including Nutritional Ketosis for the Management of Type 2 Diabetes: A 2-Year Non-randomized Clinical Trial. Front Endocrinol (Lausanne). 2019 Jun 5;10:348. doi: 10.3389/fendo.2019.00348. eCollection 2019. PMID 31231311
- [Background] Aubert G, Martin OJ, Horton JL, Lai L, Vega RB, Leone TC, Koves T, Gardell SJ, Kruger M, Hoppel CL, Lewandowski ED, Crawford PA, Muoio DM, Kelly DP. The Failing Heart Relies on Ketone Bodies as a Fuel. Circulation. 2016 Feb 23;133(8):698-705. doi: 10.1161/CIRCULATIONAHA.115.017355. Epub 2016 Jan 27. PMID 26819376
- [Background] Bertero E, Maack C. Metabolic remodelling in heart failure. Nat Rev Cardiol. 2018 Aug;15(8):457-470. doi: 10.1038/s41569-018-0044-6. PMID 29915254
- [Background] Nielsen R, Moller N, Gormsen LC, Tolbod LP, Hansson NH, Sorensen J, Harms HJ, Frokiaer J, Eiskjaer H, Jespersen NR, Mellemkjaer S, Lassen TR, Pryds K, Botker HE, Wiggers H. Cardiovascular Effects of Treatment With the Ketone Body 3-Hydroxybutyrate in Chronic Heart Failure Patients. Circulation. 2019 Apr 30;139(18):2129-2141. doi: 10.1161/CIRCULATIONAHA.118.036459. PMID 30884964
- [Background] Norwitz NG, Loh V. A Standard Lipid Panel Is Insufficient for the Care of a Patient on a High-Fat, Low-Carbohydrate Ketogenic Diet. Front Med (Lausanne). 2020 Apr 15;7:97. doi: 10.3389/fmed.2020.00097. eCollection 2020. PMID 32351962
- [Background] Soto-Mota A, Vansant H, Evans RD, Clarke K. Safety and tolerability of sustained exogenous ketosis using ketone monoester drinks for 28 days in healthy adults. Regul Toxicol Pharmacol. 2019 Dec;109:104506. doi: 10.1016/j.yrtph.2019.104506. Epub 2019 Oct 23. PMID 31655093
- [Background] Soto-Mota A, Norwitz NG, Clarke K. Why a d-beta-hydroxybutyrate monoester? Biochem Soc Trans. 2020 Feb 28;48(1):51-59. doi: 10.1042/BST20190240. PMID 32096539